CLINICAL TRIAL: NCT02263638
Title: Treatment of Refractory Hemochromatosis Rheumatism by Anakinra: a Preliminary Phase II Study
Acronym: THERA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-000609-10; 35RC13_8811_THERA (Other: Rennes University Hospital)
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Refractory Hemochromatosis Rheumatism
Keywords: hereditary haemochromatosis; rheumatism; anakinra
MeSH Terms: conditions — Hemochromatosis; Rheumatic Diseases | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anakinra (Experimental): One daily subcutaneous injection of a fixed dose of 100 mg will be administered at a fixed time by a nurse during a five day period
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — One daily subcutaneous injection of a fixed dose of 100 mg will be administered at a fixed time during a five day period

SUMMARY:
Treatment of refractory hemochromatosis rheumatism by Anakinra. Prospective, multicenter, non-randomised, single-arm, open-label, phase II trial.

DETAILED DESCRIPTION:
Hereditary hemochromatosis (HH) is a genetic disease characterized by tissue iron overload. The most common genotype is homozygosity for the p.Cys282Tyr mutation of the HFE gene (MIM 235200). It is a serious disease which can lead to life threatening complications such as cirrhosis, liver carcinoma, heart failure or diabetes mellitus. Currently, these complications can be prevented by phlebotomies. Two-thirds of patients complain of joint symptoms which represent a major cause of impaired quality of life. Phlebotomies are ineffective on HH rheumatism and patients' quality of life is very often altered while life threatening complications are prevented. Furthermore, there is a significant higher risk for joint replacement surgery in these patients compared to controls (X 9). There is currently no approved treatment for hemochromatosis rheumatism. As it looks like severe osteoarthritis, calcium pyrophosphate deposition disease (CPDD) or chondrocalcinosis, symptomatic treatments are employed such as analgesics (type I or II), non-steroidal anti-inflammatory drugs or colchicine in case of acute joint flare, corticosteroids intra-articular injections or occasionally oral glucocorticoids. However in some cases these treatments remain ineffective leading to a true disability.

Frequently, there are local inflammatory symptoms. Interleukin 1ß (IL1ß) plays a key role in the pathogenesis of crystal arthropathies (CPDD or gout).

Anakinra (IL-1Ra), a drug approved in France for rheumatoid arthritis, has been tested in short series or case controls in refractory gout, CPDD and only in two patients with HH rheumatism. The aim of this phase II study is to test the efficacy of anakinra in patients with hemochromatosis and refractory joint pain. It is also to evaluate the opportunity to perform a phase III trial. In the absence of available data on the evolution of this rheumatism treated by anakinra in this population of patients resistant to standard therapy, the investigators consider that a phase III trial would not be justifiable if the rate of success is insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age equal to or over 18 years old,
* Patients with proved hereditary hemochromatosis with homozygosity for the C282Y mutation of the HFE gene,
* Patients with rheumatism related to hemochromatosis, considered by the rheumatologist refractory to usual treatment defined by a persistent painful symptomatology despite a treatment of at least one month with level 2 analgesics (weak opioids) at maximal dose, NSAID, colchicine, steroid injection or a combination of these treatments,
* Patients with pain > 40/100mm measured by VAS (pain of the last 48 hours),
* Effective contraception to be used during treatment and until 48h after the last administration for women of reproductive age,
* Patients who have given written informed consent.

Exclusion Criteria:

* Other cause of inflammatory rheumatisms such as Rheumatoid Arthritis, Spondyloarthropathies, psoriatic arthritis, or systemic diseases,
* Ongoing treatment with Methotrexate, Hydroxychloroquine, biologic or immunosuppressive drugs
* Malignant pathology, monoclonal gammopathy,
* Intolerance to anakinra,
* Contraindications to the use of anakinra: pregnancy or breastfeeding, hypersensitivity to any of the excipients or to proteins from E. coli, severe renal impairment (creatinine clearance <30 ml / minute), neutropenia (neutrophil count <1.5 x 109 / l), ongoing infection
* Patients that cannot follow the protocol,
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Rate of patients with improvement of joint pain | Day 15
  Improvement is defined as the minimal clinically important improvement of joint pain and is assessed on a 0-100 mm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Assessment of the disease activity | Day 0, day 15, day 30, day 60, day 90
  Assessment of the disease activity by Visual analog scale (VAS)
Assessment of the number of painful joints | Day 0, day 15, day 30, day 60, day 90
  Assessment of the number of painful joints by a clinical exam
Assessment of the number of swollen joints | Day 0, day 15, day 30, day 60, day 90
  Assessment of the number of swollen joints by a clinical exam
Assessment of analgesics consumption | Day 0, day 15, day 30, day 60, day 90
Assessment of non-steroidal anti-inflammatory drugs (NSAID) consumption | Day 0, day 15, day 30, day 60, day 90
Assessment of colchicine consumption | Day 0, day 15, day 30, day 60, day 90
Assessment of steroids injections consumption | Day 0, day 15, day 30, day 60, day 90
Assessment of the quality of life | Day 0, day 15, day 30, day 90
  Assessment of the quality of life by the SF36 questionnaire
Assessment of the quality of life | Day 0, day 15, day 30, day 90
  Assessment of the quality of life by the HAQ questionnaire
Functional evaluation | Day 0, day 15, day 30, day 90
  Functional evaluation by WOMAC index for hip and knee
Functional evaluation | Day 0, day 15, day 30, day 90
  Functional evaluation by Dreiser index for hands
Assessment of joint damage | Day 0, day 90
  Assessment of joint damage by X-rays and Doppler ultrasound
Synovial fluid analysis | 3 months
  Puncture if acute joint effusion : cells count
Synovial fluid analysis | 3 months
  Puncture if acute joint effusion : search for crystals presence
Synovial fluid analysis | 3 months
  Puncture if acute joint effusion : iron parameters markers
Biological effects on inflammation and iron metabolism | Day 0, day 15, day 30, day 60, day 90
  Biological/Vaccine : iron and inflammatory markers
Time at which Cmax of anakinra was observed (Tmax) | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study
Maximum observed concentration (Cmax) of anakinra | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study
Half-life (T1/2) of anakinra | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study
Area under the concentration-time curve of time 0 to the last detectable concentration (AUC0-last) of anakinra | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study
Area under the concentration-time curve of time 0 to infinity (AUC0-∞) of anakinra | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study
Plasma clearance after administration (CL/F) of anakinra | Predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, 24 hours post-dose
  Pharmacokinetics study

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Richette, Principal Investigator — Groupe Hospitalier Lariboisière - Paris; Pascal Guggenbuhl, Principal Investigator — Rennes University Hospital
Locations (3):
- France (3):
  - CHRU de Lille, Lille
  - Groupe Hospitalier Lariboisière, Paris
  - Rennes University Hospital, Rennes